CLINICAL TRIAL: NCT03223896
Title: Pilot Study: Treatment of Gambling Disorder With Fast Acting Opiate Antagonist, Naloxone Nasal Spray
Brief Title: Treatment of Gambling Disorder With Fast Acting Opiate Antagonist, Naloxone Nasal Spray
Acronym: NALPILO
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Finnish Institute for Health and Welfare (Other Government)
Responsible Party: Principal Investigator, Hannu Alho, Research Professor, Finnish Institute for Health and Welfare
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 67016.02.01/2016
Record Dates: First submitted 2017-06-21; First posted 2017-07-21 (Actual); Last update posted 2019-09-12 (Actual); Status verified 2019-09

CONDITIONS: Gambling; Opioid; Naloxone; Spray
Keywords: antagonist; nasal
MeSH Terms: conditions — Gambling | interventions — Naloxone

STUDY DESIGN:
Intervention Model Description: Group A: max 8 mg/per day naloxone nasal spray
  Group B: max 16 mg/per day naloxone nasal spray
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Group A (Active Comparator): max 8 mg/per day naloxone nasal spray
  Interventions: Drug: Naloxone hydrochloride 20mg/ml
- Group B (Active Comparator): max 16 mg/per day naloxone nasal spray
  Interventions: Drug: Naloxone hydrochloride 20mg/ml

INTERVENTIONS:
Drug: Naloxone hydrochloride 20mg/ml — Nasal spray
  Other Names: Naloxone hyddochlodie

SUMMARY:
Non-controlled pilot study. Two groups: Group A: naloxone nasal spray max 8 mg/per day; Group B: naloxone max 16 mg/per day. Study duration 8 weeks. Brief intervention.

DETAILED DESCRIPTION:
Non-controlled pilot study. Two groups: Group A: naloxone nasal spray max 8 mg/per day; Group B: naloxone max 16 mg/per day. Study duration 8 weeks. No supportive therapy, but brief self-help booklet. Primary outcomes: adverse events, adherence and drop out analysis. Secondary outcome: gambling expenditure.

ELIGIBILITY:
Inclusion Criteria:

* age over 18 years old
* South Oaks Gambling Scale (SOGS) 5 or over points
* possibility to keep a record with phone and send text messages
* fluent in Finnish Language

Exclusion Criteria:

* active drug use (specially opioids) current use - drugs screen
* nasal abnormality or mucosal irritability
* hepatitis c virus, kidney insufficiency
* psychosis, unstable mental health, risk suicide (Beck Depression Inventory)
* pregnancy and/or breast feeding
* persons according to Finnish Medical Law 188/1999 §7-10

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2017-02-14 (Actual); Primary Completion 2017-06-30 (Actual); Study Completion 2017-06-30 (Actual)

PRIMARY OUTCOMES:
Adverse events | 8 weeks
  Diary
Adherence | 8 weeks
  Case Report Form

SECONDARY OUTCOMES:
Gambling expenditure | 8 weeks
  Money

CONTACTS AND LOCATIONS:
Overall Officials: Hannu Alho, Prof., Principal Investigator — Finnish Institute for Health and Welfare
Locations (1):
- National Institute for Heath and Welfare, Helsinki, Finland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Dowling N, Merkouris S, Lubman D, Thomas S, Bowden-Jones H, Cowlishaw S. Pharmacological interventions for the treatment of disordered and problem gambling. Cochrane Database Syst Rev. 2022 Sep 22;9(9):CD008936. doi: 10.1002/14651858.CD008936.pub2. PMID 36130734
- See also: Open accès publication on the results — https://bmjopen.bmj.com/content/9/8/e023728